CLINICAL TRIAL: NCT04430504
Title: Goal Attainment Evaluation of Multidisciplinary Telerehabilitation After Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vetrea Terveys Oy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMoK
Record Dates: First submitted 2020-05-29; First posted 2020-06-12 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Traumatic Brain Injury
Keywords: Telerehabilitation; Case series; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Case series of eligible patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (TR) (Experimental): Multidisciplinary, weekly video meetings, self-exercises at home, digital diary recordings, follow-up assessments
  Interventions: Behavioral: multidisciplinary telerehabilitation

INTERVENTIONS:
Behavioral: multidisciplinary telerehabilitation — weekly video meetings to instruct and monitor self-exercises at home

SUMMARY:
The purpose of the study is to evaluate the outcome of a multidiscplinary telerehabilitation after traumatic brain injury assessed by the patient and the therapists with respect to the overall feasibility of the therapy protocol and the effects on psychological well-being and quality of life..

DETAILED DESCRIPTION:
Patients from 18 to 60 years of age recovering after traumatic brain injury are recruited to participate in a multidisciplinary telerehabilitation containing total of 20 video meetings over a period of 4-5 months. The study design consists of a 3-day visit in rehabilitation ward for the pre-treatment clinical assessments and education on the telerehabilitation protocol. A self-exercise program is supervised and monitored using a health platform application on a tablet computer through weekly video meetings. A digital diary recordings enable the therapists to track on the progress of therapies. The primary goal is to achieve the individual goals set in the Goal Attainment Scaling. The secondary goals are related to the improvement of psychological well-being (BDI) and quality of life (WHOQOL-Bref).

ELIGIBILITY:
Inclusion Criteria:

* sequelae of traumatic brain injury
* capable of doing self exercises at home and participating in video meetings

Exclusion Criteria:

* moderate or severe aphasia
* poor recovery potential for return to school or working life based on clinical assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling | 20 weeks
  Outcome scaling: -2 (worse expected outcome), -1 (less than expected outcome), 0 (expected outcome), +1 (more than expected outcome), +2 (best expected outcome)

SECONDARY OUTCOMES:
Beck Depression Inventory | 20 weeks
  21-question inventory to yield a total score 0-63: 0-13 (no depression), 14-19 (mild depression), 20-28 (moderate depression), 29-63 (severe depression)
WHOQOL-Bref | 20 weeks
  26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items). Each domain scoring 0-100 (0 = worst, 100= best possible) to compare with age-related mean values.

CONTACTS AND LOCATIONS:
Overall Officials: Kauko Pitkänen, MD, PhD, Study Director — VetreaNeuron
Locations (1):
- VetreaNeuron, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No